CLINICAL TRIAL: NCT05855109
Title: A Prospective, Multi-national, Cross-sectional Study on a Risk-factor Guided Approach to Interstitial Lung Disease Screening in Patients With Rheumatoid Arthritis at Higher Risk for ILD Using High Resolution Computed Tomography
Brief Title: Developing a Screening Tool for Interstitial Lung Disease in People With Rheumatoid Arthritis Using Risk Factors
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0510
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Arthritis, Rheumatoid; Lung Diseases, Interstitial
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Rheumatoid Arthritis (RA): RA and 2 or more risk factors for developing Interstitial Lung Disease (ILD)

SUMMARY:
The overall aim of the study is to develop and validate a Rheumatoid Arthritis-Interstitial Lung Disease (RA-ILD) clinical prediction model (screening tool) based on risk factors to guide screening for ILD in patients with RA using High Resolution Computed Tomography (HRCT).

ELIGIBILITY:
Inclusion criteria:

1. Adult patients with RA according to 1987 American College of Rheumatology (ACR) or 2010 ACR / European League Against Rheumatism (EULAR) classification of RA, with any RA duration
2. Patient must have ≥ 2 of the following risk factors for ILD (i.e., any 2 or more):

   * Male
   * Current or previous smoker
   * Age of ≥ 60 years at RA diagnosis
   * Rheumatoid factor high-positive (titer > 3x upper limit of normal) AND/OR anti-cyclic citrullinated peptide (anti-CCP) high-positive (titer > 3x upper limit of normal) at RA diagnosis or any time after RA diagnosis
   * High/severe RA disease activity score at screening visit or within 12 months of screening visit, as defined with any of the following measures: Disease Activity Score-28 (DAS-28), Clinical Disease Activity Index (CDAI), Routine Assessment of Patient Index Data 3 (RAPID-3), Simple Disease Activity Index (SDAI), Patient Activity Scale (PAS), PAS-II
   * Presence or history of these extra-articular manifestations of RA: vasculitis, Felty's syndrome, secondary Sjogren's syndrome, cutaneous rheumatoid nodules, serositis and/or scleritis/uveitis

Exclusion criteria:

1. Patients previously diagnosed with any ILD or interstitial lung abnormality (ILA)
2. Patients who have had a chest computerized tomography (CT) in the past 2 years
3. Pregnancy at time of HRCT (to be checked in women of child-bearing potential before scan)
4. Unwilling or unable to obtain HRCT
5. Patients previously received drugs or treatments that are known to induce ILD (e.g., radiation therapy to chest region, bleomycin). Note: All disease-modifying antirheumatic drugs (DMARDs) including methotrexate and biologics are allowed.
6. Patients who have had a lung transplant
7. Patients suspected of having developed ILD due to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection / coronavirus disease 19 (COVID-19) (based on Investigators' judgement)
8. Patients diagnosed with another autoimmune disorders overlapping with RA-associated with the development of ILD (systemic sclerosis, myositis, dermatomyositis, mixed connective tissue disease, systemic lupus erythematosus, antineutrophilic cytoplasmic antibody (ANCA)-associated vasculitis or primary Sjogren's syndrome)
9. Patients currently enrolled in an investigational new drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Rheumatoid Arthritis (RA) and 2 or more risk factors for developing Interstitial Lung Disease (ILD)
Sampling Method: Probability Sample
Enrollment: 1304 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Probability score based on multi-variable diagnostic model that incorporates risk factors commonly available in clinical practice for RA-ILD screening | up to 1 year
  The endpoint of the model will be to recommend screening HRCT scan based on risk factors.
Prevalence of RA-ILD and radiological features of RA-ILD on HRCT | up to 1 year

SECONDARY OUTCOMES:
Demographics of patients with and without ILD symptoms | up to 1 year
  Age, sex, race (Baseline characteristics)
Disease characteristics of patients with and without ILD symptoms: Duration of Rheumatoid Arthritis | up to 1 year
Disease characteristics of patients with and without ILD symptoms: Disease Activity Score (DAS) 28 | up to 1 year
  The DAS28 score ranges from 0 to 9.4 with higher values reflecting a higher disease activity.
Disease characteristics of patients with and without ILD symptoms: Forced Vital Capacity | up to 1 year
Disease characteristics of patients with and without ILD symptoms: Diffusing Capacity for Carbon Monoxide | up to 1 year
Diagnostic performance of clinical prediction model in asymptomatic and symptomatic sub-populations | up to 1 year
  The overall apparent performance of the model will primarily be assessed using the Brier Score. Discrimination will be assessed using the Area Under the Curve (AUC) (c-statistic) and callibration will be analysed with a calibration plot.
Correlation of abnormal findings on pulmonary function testing (PFT) and auscultation relevant to ILD to HRCT findings | up to 1 year

CONTACTS AND LOCATIONS:
Locations (28):
- United States (5):
  - Stanford University School of Medicine, Palo Alto, California
  - University of Colorado, Aurora, Colorado
  - Harvard Medical School - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
- France (4):
  - Clinique de l'infirmerie Protestante, Caluire-et-Cuire
  - Assistance Publique - Hopitaux de Paris (AP-HP) - Hopital Cochin, Paris
  - Hopital Bichat, APHP, Paris
  - Centre Hospitalier Universitaire (CHU) de Saint-Etienne - Hopital Nord, Saint-Priest-en-Jarez
- Germany (3):
  - Rheumazentrum Prof. Dr. med Gunther Neeck, Bad Doberan
  - Charite - Universitaetsmedizin Berlin - Campus Charite Mitte (CCM), Berlin
  - Dr. Jochen Walter MD, Office Of, Rendsburg
- Italy (6):
  - Di.M.I. Irccs A.O.S.Martino (U.O.Clinica Reumatological), Genova
  - Fondazione Irccs Ca' Granda Ospedale Maggioe Policlinico Di Milano, Milan
  - Azienda Ospedaliero-Universitaria Policlinico di Modena, Modena
  - AOU di Padova, Padua
  - Fondazione Policlinico Universitario - Agostino Gemelli, Universita Cattolica del Sacro Cuore, Roma
  - Azienda Ospedaliera Universitaria Integrata di Verona - Ospedale Borgo Roma, Verona
- Spain (6):
  - Hospital Clinic de Barcelona (Hospital Clinic i Provincial), Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital General Universitario De Valencia, Valencia
  - Hospital Do Meixoeiro, Vigo
- United Kingdom (4):
  - Nottingham University Hospitals NHS Trust - Nottingham City Hospital, Nottingham
  - Southampton General Hospital - University Hospital Southampton NHS Foundation Trust, Southampton
  - Leeds University, West Yorkshire
  - Southend University Hospital - Mid Essex Hospital Services NHS Trust, Westcliff-on-Sea

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Sparks JA, Dieude P, Hoffmann-Vold AM, Burmester GR, Walsh SL, Kreuter M, Stock C, Sambevski S, Alves M, Emery P. Design of ANCHOR-RA: a multi-national cross-sectional study on screening for interstitial lung disease in patients with rheumatoid arthritis. BMC Rheumatol. 2024 May 21;8(1):19. doi: 10.1186/s41927-024-00389-4. PMID 38773593
- See also: Related Info — https://www.mystudywindow.com